CLINICAL TRIAL: NCT06466278
Title: IcoSApent ethyL to Slow Down Aortic VAlve Stenosis proGrEssion
Acronym: SALVAGE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Matthijs Boekholdt, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL81780.018.22
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medication (Experimental)
  Interventions: Drug: Icosapent ethyl
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Icosapent ethyl — 2dd2
  Arms: Medication
Drug: Placebo — 2dd2
  Arms: Placebo

SUMMARY:
This study invastigates the effect of icosapent ethyl in patients with aortic valve stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 50 years
2. Mild to moderate AVS

Exclusion Criteria:

1. Bicuspid aortic valve
2. History of chest radiotherapy
3. History of rheumatic fever
4. Moderate to severe renal failure, defined as eGFR < 30 ml/min
5. Hyperparathyroidism
6. Paget's disease
7. Diagnosis of (active) malignancy in last 5 years
8. Anticipated or planned aortic valve surgery in the next 6 months
9. Life expectancy <2 years
10. Chronic atrial fibrillation
11. Use of anticoagulant medication or dual antiplatelet therapy
12. Known hypersensitivity to fish and/or shellfish
13. Known hypersensitivity to soya
14. Malabsorption syndrome and/or chronic diarrhea
15. Women of childbearing potential who are unwilling or unable to use an acceptable method of birth control [such as oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (condoms)] to avoid pregnancy for the entire study.
16. Women who are pregnant or breastfeeding
17. Any other treatment or clinically relevant condition that could interfere with the conduct or interpretation of the study in the opinion of the investigator
18. Inability or unwillingness to comply with the protocol requirements, or deemed by investigator to be unfit for the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in aortic valve calcium (AVC) score | 2 years
  continuous variable

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No